CLINICAL TRIAL: NCT04538144
Title: Heat Waves in the Elderly: Reducing Thermal and Cardiovascular Consequences
Brief Title: Cardiovascular Responses to Heat Waves in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU_2019_1759; 1R01AG069005-01 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Aging; Hyperthermia
Keywords: aging; heat wave; cardiovascular
MeSH Terms: conditions — Hyperthermia | interventions — Hot Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Younger participants: Hot/Dry then Hot/Humid (Other): Individuals aged 18-39 years who completed the hot/dry trial first and the hot/humid trial second.
  Interventions: Other: Hot and Humid Trial; Other: Hot and Dry Trial
- Older participants: Hot/Dry then Hot/Humid (Other): Individuals aged 65 years or older who completed the hot/dry trial first and the hot/humid trial second.
  Interventions: Other: Hot and Humid Trial; Other: Hot and Dry Trial
- Younger participants: Hot/Humid then Hot/Dry (Other): Individuals aged 18-39 years who completed the hot/humid trial first and the hot/dry trial second.
  Interventions: Other: Hot and Humid Trial; Other: Hot and Dry Trial
- Older participants: Hot/Humid then Hot/Dry (Other): Individuals aged 65 years or older who completed the hot/humid trial first and the hot/dry trial second.
  Interventions: Other: Hot and Humid Trial; Other: Hot and Dry Trial

INTERVENTIONS:
Other: Hot and Humid Trial — Individuals will be exposed to a simulated heat wave (hot and humid) condition.
Other: Hot and Dry Trial — Individuals will be exposed to a simulated heat wave (hot and dry) condition.

SUMMARY:
The purpose of this study is to assess the cardiovascular responses of the elderly to heat wave conditions

DETAILED DESCRIPTION:
Heat waves are lethal and cause a disproportionate number of deaths in the elderly relative to any other age group. It is important to note that such deaths are primarily cardiovascular, not hyperthermia itself, in origin. Nevertheless, we know relatively little about the effects of aging on cardiovascular function during actual heat wave-like conditions. The central hypothesis of this work is that the elderly exhibit greater cardiovascular stress during heat wave conditions. Aim 1 will test the hypothesis that recognized impairments in thermoregulatory capacity in the elderly will culminate in heightened cardiovascular stress during prolonged exposure to heat wave conditions. Comprehensive cardiovascular and thermal responses in the elderly, relative to younger adults, will be evaluated during exposure to two prolonged heat wave conditions: hot and humid (replicating the 1995 Chicago heat wave) and very hot and dry (replicating the 2018 Los Angeles heat wave). The expected outcome from this body of work will re-shape our understanding of the consequences of aging on cardiovascular function during heat waves

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals
* 18-35 years or 65+ years of age
* Free of any underlying moderate to serious medical conditions

Exclusion Criteria:

* Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, uncontrolled hypertension, and uncontrolled hypercholesterolemia.
* Taking of any medications (such as beta blockers and non-dihydropyridine calcium channel blockers) that have known influences on either cardiac function or sweating responses.
* Abnormalities detected on routine screening.
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2
* Pregnant individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants were either screened out or withdrew before randomization.
Groups:
- Younger Participants: Hot and Humid First, Then Hot and Dry: Individuals aged 18-39 years that had the hot/humid trial first and the hot/dry trial second.
- Younger Participants: Hot and Dry First, Then Hot and Humid: Individuals aged 18-39 years that had the hot/dry trial first and the hot/humid trial second.
- Older Participants: Hot and Humid First, Then Hot and Dry: Individuals aged 65 years or older that had the hot/humid trial first and the hot/dry trial second.
- Older Participants: Hot and Dry First, Then Hot and Humid: Individuals aged 65 years or older that had the hot/dry trial first and the hot/humid trial second.
Period: First Intervention (3 Hours)
Arm/Group | Younger Participants: Hot and Humid First, Then Hot and Dry | Younger Participants: Hot and Dry First, Then Hot and Humid | Older Participants: Hot and Humid First, Then Hot and Dry | Older Participants: Hot and Dry First, Then Hot and Humid
Started | 9 | 11 | 8 | 13
Completed | 9 | 11 | 8 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Younger Participants: Hot and Humid First, Then Hot and Dry | Younger Participants: Hot and Dry First, Then Hot and Humid | Older Participants: Hot and Humid First, Then Hot and Dry | Older Participants: Hot and Dry First, Then Hot and Humid
Started | 9 | 11 | 8 | 13
Completed | 9 | 11 | 8 | 12
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Second Intervention (3 Hours)
Arm/Group | Younger Participants: Hot and Humid First, Then Hot and Dry | Younger Participants: Hot and Dry First, Then Hot and Humid | Older Participants: Hot and Humid First, Then Hot and Dry | Older Participants: Hot and Dry First, Then Hot and Humid
Started | 9 | 11 | 8 | 12
Completed | 9 | 11 | 8 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger Participants: Hot and Humid First, Then Hot and Dry | Younger Participants: Hot and Dry First, Then Hot and Humid | Older Participants: Hot and Humid First, Then Hot and Dry | Older Participants: Hot and Dry First, Then Hot and Humid | Total
Number analyzed (Participants) | 9 | 11 | 8 | 12 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6) | 29 (4) | 70 (4) | 71 (4) | 50 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 6 | 4 | 20
  Male | 5 | 5 | 2 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 8 | 10 | 7 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 6
  White | 6 | 6 | 7 | 11 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 8 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Body Temperature
Description: Core body temperature will be measured via a telemetric pill or rectal temperature probe.
Time Frame: Prior to and after the 3-hour simulated heat wave exposure.
Measure: Mean (Standard Deviation); unit: degrees Celsius (°C)
Groups:
- Younger Participants- Hot and Dry; Younger Participants: Hot and Humid: Individuals aged 18-39 years.
- Older Participants- Hot and Dry; Older Participants: Hot and Humid: Individuals aged 65 years or older.
Arm/Group | Younger Participants- Hot and Dry | Older Participants- Hot and Dry | Younger Participants: Hot and Humid | Older Participants: Hot and Humid
Number analyzed (Participants) | 20 | 20 | 20 | 20
degrees Celsius (°C) | .68 (.27) | 1.37 (.42) | .58 (.25) | 1.02 (.32)

2. Primary Outcome: Change in Peak Mitral Annular Systolic Velocity (S')
Description: Change in peak mitral annular systolic velocity was measured by tissue doppler imaging.
Time Frame: Prior to, during, and after each simulated heat wave exposure; approximately 20 min each
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Younger Participants: Hot/Dry Trial; Younger Participants: Hot/Humid Trial: Individuals aged 18-39 years.
- Older Participants: Hot/Dry Trial; Older Participants: Hot/Humid Trial: Individuals aged 65 years or older.
Arm/Group | Younger Participants: Hot/Dry Trial | Older Participants: Hot/Dry Trial | Younger Participants: Hot/Humid Trial | Older Participants: Hot/Humid Trial
Number analyzed (Participants) | 20 | 20 | 20 | 20
cm/s | 1.46 (1.54) | 3.33 (2.05) | 1.39 (1.31) | 2.09 (1.29)

3. Secondary Outcome: Ending Skin Temperature
Description: Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin.
Time Frame: At the end of the 3-hour simulated heat wave exposure.
Population: It should be noted that only 17 older participants for the hot/dry trial and 19 participants for the hot/humid trial were analyzed due to missing data/equipment issues.
Measure: Mean (Standard Deviation); unit: degrees Celsius (°C)
Arm/Group | Younger Participants: Hot/Dry Trial | Older Participants: Hot/Dry Trial | Younger Participants: Hot/Humid Trial | Older Participants: Hot/Humid Trial
Number analyzed (Participants) | 20 | 17 | 20 | 19
degrees Celsius (°C) | 37.57 (.73) | 37.37 (.85) | 36.65 (.83) | 36.05 (.58)

4. Secondary Outcome: Ending Heart Rate
Description: Heart rate will be measured via ECG electrodes attached to the participant
Time Frame: At the end of the 3-hour simulated heat wave exposure.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Younger Participants: Hot/Dry Trial | Older Participants: Hot/Dry Trial | Younger Participants: Hot/Humid Trial | Older Participants: Hot/Humid Trial
Number analyzed (Participants) | 20 | 20 | 20 | 20
beats per minute (bpm) | 82 (9) | 87 (15) | 80 (10) | 81 (14)

5. Secondary Outcome: Ending Mean Arterial Pressure
Description: Arterial blood pressure will be measured using a standard arm blood pressure cuff.
Time Frame: At the end of the 3-hour simulated heat wave exposure.
Population: It should be noted that only 19 participants were analyzed in the Hot/Humid arm because of missing data/equipment issues.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Younger Participants: Hot/Dry Trial | Older Participants: Hot/Dry Trial | Younger Participants: Hot/Humid Trial | Older Participants: Hot/Humid Trial
Number analyzed (Participants) | 20 | 20 | 20 | 19
mmHg | 77 (7) | 76 (10) | 78 (5) | 76 (8)

6. Secondary Outcome: Change in Cardiac Output
Description: Cardiac output (how much blood is ejected from the heart per minute) was measured using echocardiography.
Time Frame: Prior to and after the 3-hour simulated heat wave exposure.
Population: It should be known that only 16 participants in the hot/dry trials (younger and older) and the hot/humid trial (younger) and only 14 participants in the hot/humid trial (older) were analyzed due to missing data/equipment malfunction.
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Older Participants: Hot/Humid: Individuals aged 65 years or older.
Arm/Group | Younger Participants: Hot/Dry Trial | Older Participants: Hot/Dry Trial | Younger Participants: Hot/Humid Trial | Older Participants: Hot/Humid
Number analyzed (Participants) | 16 | 16 | 16 | 14
L/min | .88 (.77) | .75 (.82) | .38 (.52) | .76 (.96)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first consent visit to the final experimental visit of the participant. This generally encompassed a 4-week time period for each participant.
Groups:
- Younger Participants: Hot and Dry; Younger Participants: Hot and Humid: Individuals aged 18-39 years
- Older Participants: Hot and Dry; Older Participants: Hot and Humid: Individuals aged 65 years or older
Arm/Group | Younger Participants: Hot and Dry | Older Participants: Hot and Dry | Younger Participants: Hot and Humid | Older Participants: Hot and Humid
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04538144/Prot_SAP_000.pdf